CLINICAL TRIAL: NCT04393298
Title: A Phase 1/2 Open-Label, Multicenter Study to Assess the Safety, Pharmacokinetics, and Anti Tumor Activity of UCB6114 Administered Intravenously to Participants With Advanced Solid Tumors
Brief Title: A Study to Assess the Safety, Pharmacokinetics and Anti Tumor Activity of UCB6114 Administered Intravenously to Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ONC001; 2019-002598-78 (EudraCT Number)
Record Dates: First submitted 2020-03-03; First posted 2020-05-19 (Actual); Results first posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced solid tumors; UCB6114; Phase 1/2
MeSH Terms: interventions — trifluridine tipiracil drug combination; Leucovorin; Fluorouracil

STUDY DESIGN:
Intervention Model Description: Modular design, escalation & expansion modules. Depending on emerging data, not all modules may open
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A (Experimental): Study participants assigned this arm will receive UCB6114 as monotherapy in escalating cohorts at pre-specified dose levels.
  Interventions: Drug: ginisortamab
- Part A1 (Experimental): Study participants will receive predefined doses of UCB6114 as monotherapy administered intravenously at pre-specified time points.
  Interventions: Drug: ginisortamab
- Part B (Experimental): Study participants assigned to this arm will receive UCB6114 in escalating cohorts at pre-specified dose levels in combination with trifluridine/tipiracil (TFD/TPI).
  Interventions: Drug: ginisortamab; Drug: trifluridine/tipiracil
- Part C (Experimental): Study participants assigned to this arm will receive UCB6114 in escalating cohorts at pre-specified dose levels in combination with oxaliplatin, leucovorin, and 5-fluorouracil (FOLFOX) regimen.
  Interventions: Drug: ginisortamab; Drug: mFOLFOX6

INTERVENTIONS:
Drug: ginisortamab — Study participants will receive predefined doses of ginisortamab (UCB6114) administered intravenously at pre-specified time points.
  Other Names: UCB6114
Drug: trifluridine/tipiracil — Study participants will receive predefined doses of trifluridine/tipiracil (TFD/TPI) administered as film-coated tablets at pre-specified time points.
  Other Names: TAS-102; Lonsurf®
  Arms: Part B
Drug: mFOLFOX6 — Study participants will receive predefined doses of oxaliplatin, Leucovorin and 5-fluorouracil as part of the mFOLFOX6 chemotherapy regimen administered as intravenous (iv) infusion at prespecified time points.
  Other Names: Calcium folinate; 5-FU; fluorouracil
  Arms: Part C

SUMMARY:
The purpose of the study is to characterize the safety and pharmacokinetic (PK) profile of UCB6114 administered as monotherapy or in combination with selected standard of care (SOC) regimens.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 18 years of age inclusive, at the time of signing the informed consent
* Participant has advanced disease (ie, locally advanced or metastatic)
* Participant has measurable or non-measurable disease as defined by the relevant Response Evaluation Criteria in Solid Tumors (RECIST)
* Participant has an Eastern Cooperative Oncology Group (ECOG) performance status of ≤1

Part A specific:

- Participant has a histologically and/or cytologically confirmed diagnosis of one of the following advanced solid tumor types: colorectal adenocarcinoma, esophageal carcinoma, head and neck squamous cell carcinoma, lung adenocarcinoma, lung squamous cell carcinoma, pancreatic adenocarcinoma, prostate adenocarcinoma, stomach adenocarcinoma, bladder urothelial carcinoma, or breast invasive carcinoma

Part B and C specific:

- Participant has a histologically and/or cytologically confirmed diagnosis of one of the following advanced solid tumor types: colorectal adenocarcinoma, gastric adenocarcinoma, or adenocarcinoma of the gastroesophageal junction

Part A1 specific:

- Participant has histologically and/or cytologically confirmed diagnosis of one of the following advanced solid tumor types: colorectal adenocarcinoma, gastric adenocarcinoma, adenocarcinoma of the gastroesophageal junction, or pancreatic cancer

Exclusion Criteria:

* Participant has a known hypersensitivity to any components of the study medications or comparable drugs
* Active and clinically significant bacterial, fungal, or viral infection, known infections with hepatitis B, hepatitis C, known human immunodeficiency virus, or acquired immunodeficiency syndrome related illness
* Symptomatic central nervous system (CNS) malignancy or metastases. Screening of asymptomatic participants without history of CNS metastases is not required. Participants with asymptomatic CNS lesions should have completed standard therapy for their CNS lesions prior to study enrolment
* Current hematologic malignancies
* Prior organ or allogeneic stem-cell transplantation
* QT interval corrected (QTc) >450 msec
* Participant has impaired renal function
* Alanine transaminase or AST are ≥2xULN (if liver metastases are present: ≥5xULN)
* Participant has moderate or severe cardiovascular disease
* Current or chronic history of liver disease or known hepatic or biliary abnormalities other than liver metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (9):
- United States (3):
  - Onc001 50414, Los Angeles, California
  - Onc001 50470, Charleston, South Carolina
  - Onc001 50471, Houston, Texas
- United Kingdom (6):
  - Onc001 40305, Glasgow
  - Onc001 40113, London
  - Onc001 40304, Manchester
  - Onc001 40306, Newcastle upon Tyne
  - Onc001 40303, Oxford
  - Onc001 40302, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this study may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://www.Vivli.org

REFERENCES:
- [Derived] Davies GCG, Dedi N, Jones PS, Kevorkian L, McMillan D, Ottone C, Schulze MED, Scott-Tucker A, Tewari R, West S, Wright M, Rowley TF. Discovery of ginisortamab, a potent and novel anti-gremlin-1 antibody in clinical development for the treatment of cancer. MAbs. 2023 Jan-Dec;15(1):2289681. doi: 10.1080/19420862.2023.2289681. Epub 2023 Dec 12. PMID 38084840

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in July 2020 and concluded in April 2024.
Pre-assignment Details: The Participant Flow refers to the Safety Set (SS).
Groups:
- Part A: Ginisortamab 100 mg: Participants received ginisortamab monotherapy 100 milligrams (mg) as an intravenously (iv) infusion every 2 weeks (Q2W) on Day 1 and Day 15 of each 28-day treatment cycle until the occurrence of progressive disease, unacceptable toxicity, or participant withdrawal.
- Part A: Ginisortamab 250 mg: Participants received ginisortamab monotherapy 250 mg as an iv infusion Q2W on Day 1 and Day 15 of each 28-day treatment cycle until the occurrence of progressive disease, unacceptable toxicity, or participant withdrawal.
- Part A: Ginisortamab 500 mg: Participants received ginisortamab monotherapy 500 mg as an iv infusion Q2W on Day 1 and Day 15 of each 28-day treatment cycle until the occurrence of progressive disease, unacceptable toxicity, or participant withdrawal.
- Part A: Ginisortamab 1000 mg: Participants received ginisortamab monotherapy 1000 mg as an iv infusion Q2W on Day 1 and Day 15 of each 28-day treatment cycle until the occurrence of progressive disease, unacceptable toxicity, or participant withdrawal.
- Part A: Ginisortamab 2000 mg: Participants received ginisortamab monotherapy 2000 mg as an iv infusion Q2W on Day 1 and Day 15 of each 28-day treatment cycle until the occurrence of progressive disease, unacceptable toxicity, or participant withdrawal.
- Part A1: Ginisortamab 2000 mg Q2W (60-min), 28D: Participants received ginisortamab monotherapy 2000 mg as an iv infusion (60-minute infusion) Q2W on Day 1 and Day 15 of each 28-day treatment cycle until the occurrence of progressive disease, unacceptable toxicity, or participant withdrawal.
- Part A1: Ginisortamab 2000 mg Q2W (30-min), 28D: Participants received ginisortamab monotherapy 2000 mg as an iv infusion (30-minute infusion) Q2W on Day 1 and Day 15 of each 28-day treatment cycle until the occurrence of progressive disease, unacceptable toxicity, or participant withdrawal.
- Part A1: Ginisortamab 3000 mg Q3W (90-min), 21D: Participants received ginisortamab monotherapy 3000 mg as an iv infusion (90-minute infusion) every 3 weeks (Q3W) on Day 1 of each 21-day treatment cycle until the occurrence of progressive disease, unacceptable toxicity, or participant withdrawal.
- Part A1: Ginisortamab 4000 mg Q4W (120-min), 28D: Participants received ginisortamab monotherapy 4000 mg as an iv infusion (120-minute infusion) every 4 weeks (Q4W) on Day 1 of each 28-day treatment cycle until the occurrence of progressive disease, unacceptable toxicity, or participant withdrawal.
- Part B: Ginisortamab 500 mg + TFD/TPI SoC: Participants received ginisortamab 500 mg as an iv infusion Q2W in combination with orally administered trifluridine/tipiracil (TFD/TPI) on Day 1 and Day 15 of each 28-day treatment cycle until the occurrence of progressive disease, unacceptable toxicity, or participant withdrawal.
- Part B: Ginisortamab 1000 mg + TFD/TPI SoC: Participants received ginisortamab 1000 mg as an iv infusion Q2W in combination with orally administered TFD/TPI on Day 1 and Day 15 of each 28-day treatment cycle until the occurrence of progressive disease, unacceptable toxicity, or participant withdrawal.
- Part B: Ginisortamab 2000 mg + TFD/TPI SoC: Participants received ginisortamab 2000 mg as an iv infusion Q2W in combination with orally administered TFD/TPI on Day 1 and Day 15 of each 28-day treatment cycle until the occurrence of progressive disease, unacceptable toxicity, or participant withdrawal.
- Part C: Ginisortamab 500 mg + mFOLFOX6 SoC: Participants received ginisortamab 500 mg as an iv infusion Q2W in combination with mFOLFOX6 chemotherapy (oxaliplatin, leucovorin, and 5-fluorouracil) on Day 1 and Day 15 of each 28-day treatment cycle until the occurrence of progressive disease, unacceptable toxicity, or participant withdrawal.
- Part C: Ginisortamab 1000 mg + mFOLFOX6 SoC: Participants received ginisortamab 1000 mg as an iv infusion Q2W in combination with mFOLFOX6 chemotherapy (oxaliplatin, leucovorin, and 5-fluorouracil) on Day 1 and Day 15 of each 28-day treatment cycle until the occurrence of progressive disease, unacceptable toxicity, or participant withdrawal.
- Part C: Ginisortamab 2000 mg + mFOLFOX6 SoC: Participants received ginisortamab 2000 mg as an iv infusion Q2W in combination with mFOLFOX6 chemotherapy (oxaliplatin, leucovorin, and 5-fluorouracil) on Day 1 and Day 15 of each 28-day treatment cycle until the occurrence of progressive disease, unacceptable toxicity, or participant withdrawal.
Period: Overall Study
Arm/Group | Part A: Ginisortamab 100 mg | Part A: Ginisortamab 250 mg | Part A: Ginisortamab 500 mg | Part A: Ginisortamab 1000 mg | Part A: Ginisortamab 2000 mg | Part A1: Ginisortamab 2000 mg Q2W (60-min), 28D | Part A1: Ginisortamab 2000 mg Q2W (30-min), 28D | Part A1: Ginisortamab 3000 mg Q3W (90-min), 21D | Part A1: Ginisortamab 4000 mg Q4W (120-min), 28D | Part B: Ginisortamab 500 mg + TFD/TPI SoC | Part B: Ginisortamab 1000 mg + TFD/TPI SoC | Part B: Ginisortamab 2000 mg + TFD/TPI SoC | Part C: Ginisortamab 500 mg + mFOLFOX6 SoC | Part C: Ginisortamab 1000 mg + mFOLFOX6 SoC | Part C: Ginisortamab 2000 mg + mFOLFOX6 SoC
Started | 3 | 5 | 5 | 6 | 6 | 8 | 8 | 8 | 8 | 9 | 4 | 8 | 5 | 3 | 7
Completed | 1 | 1 | 2 | 3 | 3 | 1 | 4 | 5 | 2 | 5 | 3 | 3 | 3 | 2 | 0
Not Completed | 2 | 4 | 3 | 3 | 3 | 7 | 4 | 3 | 6 | 4 | 1 | 5 | 2 | 1 | 7
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Consent withdrawn by participant, not due to AE | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Progression | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Passed Away on The 30 Oct 2020 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Disease Progression Confirmed by Scans (CT/MRI) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Clinical Progression | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Disease Progression | 0 | 1 | 0 | 0 | 0 | 3 | 2 | 1 | 2 | 1 | 0 | 3 | 0 | 0 | 1
Not completed — Since no Treatment Administered at Cycle 2 Day 15 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Further Deterioration Noted at Clinic review | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease (PD) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Started a New Cancer Treatment | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor decision- sepsis (treatment delay) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Due to symptoms (New Brain Metastases) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Clinical Progression: Not suitable for SFU return | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1
Not completed — Progressive Disease - New Brain Mets on CT Head | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease and Subsequent Death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Patient Passed Away | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Patient Deceased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Patient Discharged to Hospice | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Symptomatic Cancer - Unfit to take a call | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Clinical Progression in Combination with AE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set (SS) which consisted of all study participants who received at least 1 full or partial dose of Ginisortamab (UCB6114).
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Ginisortamab 100 mg | Part A: Ginisortamab 250 mg | Part A: Ginisortamab 500 mg | Part A: Ginisortamab 1000 mg | Part A: Ginisortamab 2000 mg | Part A1: Ginisortamab 2000 mg Q2W (60-min), 28D | Part A1: Ginisortamab 2000 mg Q2W (30-min), 28D | Part A1: Ginisortamab 3000 mg Q3W (90-min), 21D | Part A1: Ginisortamab 4000 mg Q4W (120-min), 28D | Part B: Ginisortamab 500 mg + TFD/TPI SoC | Part B: Ginisortamab 1000 mg + TFD/TPI SoC | Part B: Ginisortamab 2000 mg + TFD/TPI SoC | Part C: Ginisortamab 500 mg + mFOLFOX6 SoC | Part C: Ginisortamab 1000 mg + mFOLFOX6 SoC | Part C: Ginisortamab 2000 mg + mFOLFOX6 SoC | Total
Number analyzed (Participants) | 3 | 5 | 5 | 6 | 6 | 8 | 8 | 8 | 8 | 9 | 4 | 8 | 5 | 3 | 7 | 93
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.0 (1.0) | 54.4 (11.0) | 58.2 (12.2) | 65.3 (8.0) | 60.7 (9.5) | 56.6 (12.0) | 67.3 (6.3) | 60.9 (6.7) | 60.8 (17.6) | 57.6 (9.5) | 51.5 (6.2) | 57.6 (14.2) | 58.6 (10.7) | 63.0 (13.0) | 61.1 (9.1) | 59.9 (10.7)
Age, Customized [Count of Participants; unit: Participants]
  18 - <65 years | 1 | 4 | 3 | 3 | 3 | 7 | 3 | 5 | 4 | 7 | 4 | 7 | 3 | 2 | 5 | 61
  65 - <85 years | 2 | 1 | 2 | 3 | 3 | 1 | 5 | 3 | 4 | 2 | 0 | 1 | 2 | 1 | 2 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 3 | 2 | 1 | 3 | 3 | 5 | 2 | 4 | 2 | 2 | 2 | 1 | 3 | 35
  Male | 3 | 3 | 2 | 4 | 5 | 5 | 5 | 3 | 6 | 5 | 2 | 6 | 3 | 2 | 4 | 58
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 4
  Black or African American | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 0 | 6
  White | 3 | 4 | 4 | 6 | 6 | 8 | 8 | 8 | 8 | 6 | 3 | 8 | 4 | 1 | 5 | 82
  Other/Mixed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 3 | 5 | 5 | 6 | 6 | 8 | 8 | 8 | 8 | 9 | 4 | 8 | 5 | 3 | 7 | 93

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study medication, whether or not considered related to the study medication. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study medication. A treatment-emergent adverse event (TEAE) was defined as any AE with a start date on or after the first dose of UCB6114 up until the last dose of Ginisortamab (UCB6114) +30 days (i.e. up to 3.8 years).
Time Frame: From Baseline until the End of Study (up to 3.8 years)
Population: The SS consisted of all study participants who received at least 1 full or partial dose of Ginisortamab (UCB6114).
Measure: Number; unit: percentage of participants
Arm/Group | Part A: Ginisortamab 100 mg | Part A: Ginisortamab 250 mg | Part A: Ginisortamab 500 mg | Part A: Ginisortamab 1000 mg | Part A: Ginisortamab 2000 mg | Part A1: Ginisortamab 2000 mg Q2W (60-min), 28D | Part A1: Ginisortamab 2000 mg Q2W (30-min), 28D | Part A1: Ginisortamab 3000 mg Q3W (90-min), 21D | Part A1: Ginisortamab 4000 mg Q4W (120-min), 28D | Part B: Ginisortamab 500 mg + TFD/TPI SoC | Part B: Ginisortamab 1000 mg + TFD/TPI SoC | Part B: Ginisortamab 2000 mg + TFD/TPI SoC | Part C: Ginisortamab 500 mg + mFOLFOX6 SoC | Part C: Ginisortamab 1000 mg + mFOLFOX6 SoC | Part C: Ginisortamab 2000 mg + mFOLFOX6 SoC
Number analyzed (Participants) | 3 | 5 | 5 | 6 | 6 | 8 | 8 | 8 | 8 | 9 | 4 | 8 | 5 | 3 | 7
percentage of participants | 100 | 100 | 100 | 100 | 100 | 87.5 | 100 | 87.5 | 100 | 100 | 100 | 100 | 100 | 100 | 100

2. Primary Outcome: Percentage of Participants Based on Severity of Treatment-emergent Adverse Events
Description: AE is any untoward medical occurrence in patient or clinical study participant, temporally associated with use of study medication, whether or not considered related to study medication. AE can therefore be any unfavorable and unintended sign (including abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with use of study medication. TEAE: any AE with start date on or after first dose of UCB6114 up until last dose of Ginisortamab(UCB6114)+30 days. Event for which no Common Terminology Criteria for AE (CTCAE) severity grade was recorded by investigator but intensity was recorded instead was assigned as follows to CTCAE severity grade:Severe=Grade 3, Life Threatening (indicated on electronic case report form (eCRF) for event that is serious)=Grade 4, Death (indicated on the eCRF for event that is serious or has outcome of death)=Grade 5. As planned, data reported for National Cancer Institute (NCI) CTCAE grade >=3 TEAEs and related TEAEs.
Time Frame: From Baseline until the End of Study (up to 3.8 years)
Population: The SS consisted of all study participants who received at least 1 full or partial dose of Ginisortamab (UCB6114).
Measure: Number; unit: percentage of participants
Arm/Group | Part A: Ginisortamab 100 mg | Part A: Ginisortamab 250 mg | Part A: Ginisortamab 500 mg | Part A: Ginisortamab 1000 mg | Part A: Ginisortamab 2000 mg | Part A1: Ginisortamab 2000 mg Q2W (60-min), 28D | Part A1: Ginisortamab 2000 mg Q2W (30-min), 28D | Part A1: Ginisortamab 3000 mg Q3W (90-min), 21D | Part A1: Ginisortamab 4000 mg Q4W (120-min), 28D | Part B: Ginisortamab 500 mg + TFD/TPI SoC | Part B: Ginisortamab 1000 mg + TFD/TPI SoC | Part B: Ginisortamab 2000 mg + TFD/TPI SoC | Part C: Ginisortamab 500 mg + mFOLFOX6 SoC | Part C: Ginisortamab 1000 mg + mFOLFOX6 SoC | Part C: Ginisortamab 2000 mg + mFOLFOX6 SoC
Number analyzed (Participants) | 3 | 5 | 5 | 6 | 6 | 8 | 8 | 8 | 8 | 9 | 4 | 8 | 5 | 3 | 7
percentage of participants
  NCI CTCAE grade >=3 TEAEs | 66.7 | 40.0 | 40.0 | 0 | 50.0 | 62.5 | 50.0 | 37.5 | 62.5 | 55.6 | 75.0 | 87.5 | 100 | 100 | 85.7
  NCI CTCAE grade >=3 related TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12.5 | 22.2 | 0 | 25.0 | 40.0 | 0 | 14.3

3. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: DLT defined as any AE at least related to study medication that occurs during Cycle 1 and met following criteria: Grade (Gr) 3 or 4 nonhematological toxicity according to NCI CTCAE (Version 5.0) except for alopecia, or nausea, vomiting, or diarrhea that reverses to Gr ≤2 within 24 hours (hr) with appropriate medical therapy; Gr 3 or 4 biochemical abnormality that persists despite maximal supportive treatment or biochemical abnormalities that is symptomatic and nontransient; Any Gr ≥3 hematological toxicity of >5 days duration or febrile neutropenia (absolute neutrophil count [ANC]<1000/cubic millimeter[mm3] with single temperature of >38.3°C or sustained temperature ≥38°C for more than one hr), infection with Gr 3 or 4 neutropenia, thrombocytopenia with bleeding or requiring platelet transfusion, or Gr 4 thrombocytopenia; Prolonged Gr 2 diarrhea (>7 days) despite adequate antidiarrheal medication, or multiple Grade 1or 2 toxicities(eg, Gr 1 or 2 diarrhea, vomiting, rash, and fatigue).
Time Frame: From Baseline throughout 28 days (Cycle 1)
Population: The SS consisted of all study participants who received at least 1 full or partial dose of Ginisortamab (UCB6114).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Ginisortamab 100 mg | Part A: Ginisortamab 250 mg | Part A: Ginisortamab 500 mg | Part A: Ginisortamab 1000 mg | Part A: Ginisortamab 2000 mg | Part A1: Ginisortamab 2000 mg Q2W (60-min), 28D | Part A1: Ginisortamab 2000 mg Q2W (30-min), 28D | Part A1: Ginisortamab 3000 mg Q3W (90-min), 21D | Part A1: Ginisortamab 4000 mg Q4W (120-min), 28D | Part B: Ginisortamab 500 mg + TFD/TPI SoC | Part B: Ginisortamab 1000 mg + TFD/TPI SoC | Part B: Ginisortamab 2000 mg + TFD/TPI SoC | Part C: Ginisortamab 500 mg + mFOLFOX6 SoC | Part C: Ginisortamab 1000 mg + mFOLFOX6 SoC | Part C: Ginisortamab 2000 mg + mFOLFOX6 SoC
Number analyzed (Participants) | 3 | 5 | 5 | 6 | 6 | 8 | 8 | 8 | 8 | 9 | 4 | 8 | 5 | 3 | 7
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0

4. Secondary Outcome: Part A and A1: UCB6114 Serum Concentration by Scheduled Assessment and Cohort
Description: Blood samples for ginisortamab serum concentration analysis were collected at different timepoints following the first dose of ginisortamab. The data is reported for Part A and A1. Pharmacokinetic Set (PKS). Lower Limit of Quantitation (LLOQ).
Time Frame: Parts A: Cycle 1 (Day 1 end of infusion [EOI] and Day 15 Predose), Cycle 2 (Day 1 Predose and Day 15 Predose); Part A 1: Cycle 1 (Day 1 EOI and Day 15 Predose), Cycle 2 (Day 1 Predose)
Population: PKS:all participants of SS with >=1 evaluable PKS concentration (ie, sample above LLOQ[0.02μg/mL] and for which date, sample time, prior date dosing time are known). Number analyzed:participants evaluable at specified time points. Dosing was only performed on Day 1 of each cycle for Part A1:Ginisortamab 3000mg Q3W(90-min) 21-day and Ginisortamab 4000mg Q4W(120-min) 28-day arms. Hence, Predose, Day 15 of Cycle 1 was not collected. No arms of Part A1 had data collection on Cycle 2 Day 15 Predose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (ug/mL)
Arm/Group | Part A: Ginisortamab 100 mg | Part A: Ginisortamab 250 mg | Part A: Ginisortamab 500 mg | Part A: Ginisortamab 1000 mg | Part A: Ginisortamab 2000 mg | Part A1: Ginisortamab 2000 mg Q2W (60-min), 28D | Part A1: Ginisortamab 2000 mg Q2W (30-min), 28D | Part A1: Ginisortamab 3000 mg Q3W (90-min), 21D | Part A1: Ginisortamab 4000 mg Q4W (120-min), 28D
Number analyzed (Participants) | 3 | 5 | 5 | 6 | 6 | 8 | 8 | 8 | 8
microgram per milliliter (ug/mL)
  Cycle 1 Day 1 EOI: number analyzed (Participants) | 3 | 5 | 4 | 5 | 6 | 8 | 8 | 8 | 5
  Cycle 1 Day 1 EOI | 18.0477 (10.0206) | 72.5261 (24.1924) | 130.7757 (14.1088) | 277.5536 (10.8287) | 552.3530 (19.5548) | 592.2331 (26.1556) | 593.1846 (22.2154) | 946.0883 (19.3798) | 1357.6103 (20.4135)
  Cycle 1 Day 15 Predose: number analyzed (Participants) | 3 | 5 | 5 | 6 | 5 | 7 | 8 | 0 | 0
  Cycle 1 Day 15 Predose | 4.4210 (10.1288) | 12.8115 (27.1385) | 24.3743 (31.2011) | 61.4527 (33.1491) | 92.0396 (38.4595) | 105.5277 (25.1756) | 97.1957 (39.3439) |  |
  Cycle 2 Day 1 Predose: number analyzed (Participants) | 2 | 1 | 5 | 6 | 4 | 4 | 8 | 6 | 7
  Cycle 2 Day 1 Predose | NA (NA) — GeoMean and GeoCV (%) were only calculated if at least 2/3 of the concentrations are quantified at the respective timepoint. | NA (NA) — GeoMean and GeoCV (%) were only calculated if at least 2/3 of the concentrations are quantified at the respective timepoint. | 34.6409 (26.9986) | 67.0799 (37.9557) | 149.3886 (37.0769) | 193.4242 (34.5942) | 147.2154 (26.4979) | 124.7274 (44.3198) | 98.9331 (33.8567)
  Cycle 2 Day 15 Predose: number analyzed (Participants) | 1 | 1 | 4 | 5 | 4 | 0 | 0 | 0 | 0
  Cycle 2 Day 15 Predose | NA (NA) — GeoMean and GeoCV (%) were only calculated if at least 2/3 of the concentrations are quantified at the respective timepoint. | NA (NA) — GeoMean and GeoCV (%) were only calculated if at least 2/3 of the concentrations are quantified at the respective timepoint. | 42.6861 (38.1929) | 78.2336 (35.0467) | 166.4011 (34.1041) |  |  |  |

5. Secondary Outcome: Part B and C: UCB6114 Concentration by Scheduled Assessment and Dose Level
Description: Blood samples for ginisortamab serum concentration analysis were collected at timepoints following (Cycle 1 Day 1) and the (Cycle 2 Day 1) administration of ginisortamab. Data is reported for Part B and Part C.
Time Frame: Part B and C: Cycle 1 (Day 1 EOI and Day 15 Predose), Cycle 2 (Day 1 Predose and Day 15 Predose)
Population: The PKS included all study participants in the SS (all study participants who received at least 1 full or partial dose of Ginisortamab [UCB6114]) who had at least 1 evaluable PKS concentration (ie, a sample which is above the lower limit of quantitation [0.02μg/mL] and for which the date and time of the sample and prior date and time of dosing are known). Here, number analyzed signifies participants who were evaluable at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part B: Ginisortamab 500 mg + TFD/TPI SoC | Part B: Ginisortamab 1000 mg + TFD/TPI SoC | Part B: Ginisortamab 2000 mg + TFD/TPI SoC | Part C: Ginisortamab 500 mg + mFOLFOX6 SoC | Part C: Ginisortamab 1000 mg + mFOLFOX6 SoC | Part C: Ginisortamab 2000 mg + mFOLFOX6 SoC
Number analyzed (Participants) | 9 | 4 | 8 | 5 | 3 | 7
ug/mL
  Cycle 1 Day 1 EOI: number analyzed (Participants) | 7 | 4 | 7 | 5 | 3 | 7
  Cycle 1 Day 1 EOI | 104.0606 (15.3565) | 250.8708 (7.6032) | 463.5265 (28.6333) | 122.8221 (14.8778) | 175.0745 (34.7390) | 471.9576 (17.1727)
  Cycle 1 Day 15 Predose: number analyzed (Participants) | 8 | 3 | 7 | 5 | 3 | 7
  Cycle 1 Day 15 Predose | 19.7473 (42.6072) | 37.4171 (14.8496) | 83.4236 (30.8533) | 16.8917 (33.2664) | 32.3094 (56.2327) | 70.7026 (50.9842)
  Cycle 2 Day 1 Predose: number analyzed (Participants) | 6 | 3 | 6 | 5 | 3 | 5
  Cycle 2 Day 1 Predose | 33.0061 (35.3957) | 61.0398 (5.0117) | 118.0926 (29.3051) | 25.4863 (53.6347) | 82.7657 (47.9648) | 141.6084 (30.8310)
  Cycle 2 Day 15 Predose: number analyzed (Participants) | 6 | 4 | 5 | 3 | 2 | 3
  Cycle 2 Day 15 Predose | 38.3595 (42.1013) | 55.0249 (39.4082) | 135.5849 (32.8644) | 24.7120 (83.6183) | NA (NA) — GeoMean and GeoCV (%) were only calculated if at least 2/3 of the concentrations are quantified at the respective timepoint. | 135.0042 (43.8716)

ADVERSE EVENTS:
Time Frame: From Baseline up to End of the Study (up to 3.8 years)
Description: A TEAE was defined as any AE with a start date on or after the first dose of UCB6114 until the last dose of Ginisortamab (UCB6114) +30 days. A pre-treatment AE which increased in severity on or after the first dose of study treatment was also counted as a TEAE. The SS consisted of all study participants who received at least 1 full or partial dose of Ginisortamab (UCB6114).
Arm/Group | Part A: Ginisortamab 100 mg | Part A: Ginisortamab 250 mg | Part A: Ginisortamab 500 mg | Part A: Ginisortamab 1000 mg | Part A: Ginisortamab 2000 mg | Part A1: Ginisortamab 2000 mg Q2W (60-min), 28D | Part A1: Ginisortamab 2000 mg Q2W (30-min), 28D | Part A1: Ginisortamab 3000 mg Q3W (90-min), 21D | Part A1: Ginisortamab 4000 mg Q4W (120-min), 28D | Part B: Ginisortamab 500 mg + TFD/TPI SoC | Part B: Ginisortamab 1000 mg + TFD/TPI SoC | Part B: Ginisortamab 2000 mg + TFD/TPI SoC | Part C: Ginisortamab 500 mg + mFOLFOX6 SoC | Part C: Ginisortamab 1000 mg + mFOLFOX6 SoC | Part C: Ginisortamab 2000 mg + mFOLFOX6 SoC
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/5 | 0/5 | 0/6 | 0/6 | 0/8 | 0/8 | 0/8 | 1/8 | 0/9 | 0/4 | 0/8 | 0/5 | 1/3 | 1/7
Serious Adverse Events (participants affected / at risk) | 2/3 | 3/5 | 1/5 | 0/6 | 1/6 | 1/8 | 2/8 | 2/8 | 5/8 | 4/9 | 2/4 | 4/8 | 5/5 | 1/3 | 2/7
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 5/5 | 6/6 | 6/6 | 7/8 | 8/8 | 7/8 | 8/8 | 9/9 | 4/4 | 8/8 | 5/5 | 3/3 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Ginisortamab 100 mg (N=3) | Part A: Ginisortamab 250 mg (N=5) | Part A: Ginisortamab 500 mg (N=5) | Part A: Ginisortamab 1000 mg (N=6) | Part A: Ginisortamab 2000 mg (N=6) | Part A1: Ginisortamab 2000 mg Q2W (60-min), 28D (N=8) | Part A1: Ginisortamab 2000 mg Q2W (30-min), 28D (N=8) | Part A1: Ginisortamab 3000 mg Q3W (90-min), 21D (N=8) | Part A1: Ginisortamab 4000 mg Q4W (120-min), 28D (N=8) | Part B: Ginisortamab 500 mg + TFD/TPI SoC (N=9) | Part B: Ginisortamab 1000 mg + TFD/TPI SoC (N=4) | Part B: Ginisortamab 2000 mg + TFD/TPI SoC (N=8) | Part C: Ginisortamab 500 mg + mFOLFOX6 SoC (N=5) | Part C: Ginisortamab 1000 mg + mFOLFOX6 SoC (N=3) | Part C: Ginisortamab 2000 mg + mFOLFOX6 SoC (N=7)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urogenital fistula (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (3) | 1 (2) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site thrombosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Ginisortamab 100 mg (N=3) | Part A: Ginisortamab 250 mg (N=5) | Part A: Ginisortamab 500 mg (N=5) | Part A: Ginisortamab 1000 mg (N=6) | Part A: Ginisortamab 2000 mg (N=6) | Part A1: Ginisortamab 2000 mg Q2W (60-min), 28D (N=8) | Part A1: Ginisortamab 2000 mg Q2W (30-min), 28D (N=8) | Part A1: Ginisortamab 3000 mg Q3W (90-min), 21D (N=8) | Part A1: Ginisortamab 4000 mg Q4W (120-min), 28D (N=8) | Part B: Ginisortamab 500 mg + TFD/TPI SoC (N=9) | Part B: Ginisortamab 1000 mg + TFD/TPI SoC (N=4) | Part B: Ginisortamab 2000 mg + TFD/TPI SoC (N=8) | Part C: Ginisortamab 500 mg + mFOLFOX6 SoC (N=5) | Part C: Ginisortamab 1000 mg + mFOLFOX6 SoC (N=3) | Part C: Ginisortamab 2000 mg + mFOLFOX6 SoC (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 1 (2) | 2 (5) | 5 (12) | 1 (2) | 6 (14) | 3 (11) | 1 (5) | 2 (4)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (14) | 3 (17) | 3 (8) | 1 (1) | 1 (3) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 2 (2) | 1 (3) | 1 (1) | 1 (2)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 2 (4) | 1 (1) | 1 (2) | 0 (0) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aorto-oesophageal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 4 (4) | 3 (3) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (7) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 3 (6) | 2 (2) | 2 (2) | 3 (4) | 2 (3) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 2 (2) | 2 (2) | 1 (3) | 4 (4) | 1 (1) | 2 (3) | 2 (3) | 1 (2) | 6 (12) | 2 (3) | 4 (6) | 5 (5) | 0 (0) | 4 (4)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 5 (6) | 2 (2) | 1 (1) | 4 (7) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (2) | 1 (1) | 3 (3) | 3 (8) | 2 (4) | 3 (4) | 5 (6) | 0 (0) | 3 (4) | 5 (8) | 2 (2) | 2 (3) | 2 (3) | 1 (2) | 5 (6)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Craniofacial fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 3 (3) | 2 (4) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 1 (1) | 2 (5) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram T wave amplitude decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (5) | 1 (1) | 2 (4) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 4 (7) | 1 (1) | 0 (0) | 3 (4)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (11) | 1 (2) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 6 (7) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 1 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (2)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Neurotoxicity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 0 (0)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydroureter (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/98/NCT04393298/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-13): https://cdn.clinicaltrials.gov/large-docs/98/NCT04393298/SAP_001.pdf